CLINICAL TRIAL: NCT01554995
Title: A Phase I Clinical Study, Randomized, Double-blind, Placebo-controlled, Single Dose, Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LCB01-0371 in Healthy Male Subjects
Brief Title: A Clinical Study, Randomized, Double-blind, Placebo-controlled, Single Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCB01-0371-11-1-01
Record Dates: First submitted 2012-03-09; First posted 2012-03-15 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: LCB01-0371
MeSH Terms: interventions — delpazolid; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCB01-0371 (Experimental): active
  Interventions: Drug: LCB01-0371
- Linezolid (Experimental): comparator
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: LCB01-0371 — LCB01-0371 50mg (Cohort 1) 100mg (Cohort 2) 200mg (Cohort 3) 400mg (Cohort 4) 600mg (Cohort 5)
  Arms: LCB01-0371
Drug: Linezolid — Linezolid 600 mg (Cohort 9) none
  Arms: Linezolid

SUMMARY:
Primary

- To investigate the safety and tolerability of LCB01-0371 after a single oral dose

Secondary

* To investigate the pharmacokinetic characteristics of LCB01-0371 after a single oral dose
* To investigate the safety of LCB01-0371 after a single oral dose

DETAILED DESCRIPTION:
* To investigate the pharmacokinetic characteristics of LCB01-0371 after a single oral dose
* To investigate the safety of LCB01-0371 after a single oral dose

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Male between 20 and 45 years of age at the time of screening
2. Subjects with body mass index (BMI) between 20 and 27 at the time of screening
3. Agree to continue to use a medically reliable dual contraception and not to donate sperm until 30th days of study completion
4. Capable of giving written informed consent, willing to participate in this clinical trial, and willing to comply with all study requirements

Exclusion Criteria:

1. History of liver, kidney, respiratory, musculoskeletal, endocrinologic, neuropsychiatric, hemato-oncologic, or cardiovascular problem(s).
2. History of gastrointestinal problem (e.g. Crohn's disease, gastro-intestinal ulcer) which is affect to absorption within 6 months from screening
3. History of hypersensitivity or clinically significant adverse drug reaction(s) to the LCB01-0371, same class of the study drugs (linezolid), or other drugs including aspirin and antibiotics.
4. History of drug abuse or positive result at urine drug screening test
5. AST, ALT, r-GT, billirubin(total) values over than 1.5 times of ULN

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 7 days
  Summary statistics for SAD parts will be prepared for measured values and changes from baseline values for each dose group. Placebo subjects will serve as the control. Summaries of treatment-emergent and clinically important abnormalities in ECG, physical examination, vital signs, and laboratory (clinical chemistry, hematology, coagulation, urinalysis) data will be provided. The incidence of adverse events(AEs) will be tabulated and compared across dose group in the SAD parts.

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph. D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho YS, Lim HS, Lee SH, Cho YL, Nam HS, Bae KS. Pharmacokinetics, Pharmacodynamics, and Tolerability of Single-Dose Oral LCB01-0371, a Novel Oxazolidinone with Broad-Spectrum Activity, in Healthy Volunteers. Antimicrob Agents Chemother. 2018 Jun 26;62(7):e00451-18. doi: 10.1128/AAC.00451-18. Print 2018 Jul. PMID 29712654